CLINICAL TRIAL: NCT02079077
Title: Limiting HIV Target Cells by Inducing Immune Quiescence in the Female Genital Tract
Brief Title: Inducing Immune Quiescence to Prevent HIV Infection in Women
Acronym: IIQ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: University of Nairobi (Other)
Responsible Party: Principal Investigator, Dr. Keith Fowke, Professor Department of Medical Microbiology, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: B2013:042; MOP#86721 (Other Grant/Funding Number: Canadian Institue of Health Research); S5-0386-01 (Other Grant/Funding Number: Grand Challenge Canada)
Record Dates: First submitted 2014-03-03; First posted 2014-03-05 (Estimated); Results first posted 2019-10-10 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-09

CONDITIONS: HIV
Keywords: HIV, Immune quiescence, ASA, Hydroxychloroquin
MeSH Terms: interventions — Aspirin; Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acetylsalicylic Acid (ASA) (Other): ASA 81 mg. p.o. daily for two months
  Interventions: Drug: Acetylsalicylic Acid (ASA)
- Hydroxychloroquine (HCQ) (Other): Hydroxychloroquine (HCQ) 200 mg. o.d. p.o. for two months.
  Interventions: Drug: Hydroxychloroquine (HCQ)

INTERVENTIONS:
Drug: Acetylsalicylic Acid (ASA) — Acetylsalicylic Acid (ASA) 81 mg. oral daily for two months
  Arms: Acetylsalicylic Acid (ASA)
Drug: Hydroxychloroquine (HCQ) — Hydroxychloroquine (HCQ) 200 mg. oral, daily for two months.
  Arms: Hydroxychloroquine (HCQ)

SUMMARY:
In this project, the investigators want to analyse the capacity of Acetylsalicylic acid and hydoxychlroquin (HCQ) to induce an Immune Quiescence (IQ) phenotype, which has been previously associated with natural protection to HIV infection. This phenotype is characterized by lower expression of genes involved in cellular activation, lower resting levels of inflammatory cytokine production, lower level of systemic activated T cells, increased levels of systemic T regulatory, increased production of anti-viral anti-protease serpins at the female genital tract and reduced numbers of HIV target cells (mainly CD4+ CCR5+ T cells) in the FGT ( female genital tract).

The objective of this study is to determine if daily oral administration of Acetylsalicylic acid or hydroxychlroroquin can reduce systemic and mucosal immune activation in HIV negative women.

DETAILED DESCRIPTION:
The investigators will enrol 80 non female sex work low-risk HIV negative women and 80 HIV negative female sex worker HIV negative form Nairobi, Kenya and followed for a 3 months period.

During the first month, samples will be taken on a monthly basis

* blood,
* vaginal samples: cytobrush/scarper and cervico vaginal lavage (CVL). This is done to determine the baseline levels of systemic and mucosal immune activation of each woman. In this way, every women is acting as her own control thereby reducing variation between control and participant.

Chemokine/cytokine level, as well as cellular immune activation and T regulatory cells will be assessed.

At month two: the women will be divided in two different arms (oral administration of hydroxychloroquine: 200mg/day or Acetylsalicylic acid 81mg/day) and followed, on a monthly basis, for an 8 additional weeks.

During this time, monthly blood and vaginal samples (cytobrush/scraper and CVL) the investigators will be taken. They will measure change in the systemic and mucosal immune activation.

Immune Quiescence phenotype (decrease of T cells immune activation, lower immune genes activation expression and pro-inflammatory cytokine/chemokine expression) will be evaluated by flow cytometry, microarray, and multiplex bead array technology.

Here is how samples will be taken:

1. A sample of cervical mucus will be collected by using a cotton swab rotated 360º in the cervical os, and a second swab used to collect secretions from the posterior vaginal fornix. Both swabs will be transferred into a single vial containing 5 mL of phosphate-buffered saline (PBS) which will be transported to the laboratory to be tested and cultured for sexually transmitted infections such as gonorrhea, chlamydia etc.
2. Cervical cells will be collected by using a small brush and a wooden spatula. Both specimen will be transferred into a 15ml conical tube containing 5 ml of PBS. This specimen will be used to characterize the cellular populations in the specimen.
3. Cervico vaginal lavage will be performed by washing the endocervix with 2 ml of sterile 1x PBS. The liquid will be collected form the posterior fornix. Samples will be placed into a conical tube, centrifuged to remove cellular debris and the supernatant will be stored at -70°C and will be shipped in liquid nitrogen dry shipper to Winnipeg, Manitoba. Those specimens will be used for innate soluble factor detection (chemokines, cytokines, antibodies, innate protein, etc
4. 30ml of venous blood will be taken. (Peripheral Blood Mononuclear Cells will be extracted for immune activation analysis, DNA will be used for immune genes expression, plasma will be used for protein and innate soluble factor detection.)

   .

ELIGIBILITY:
Inclusion criteria:

1. Age greater than 18 years old and less than 50 years old
2. Uterus and cervix present
3. Willing to take daily acetylsalicylic acid or HCQ
4. Willing to undergo pelvic exams
5. In general good health, no chronic infection and not taking any anti-inflammatory or immunosuppressors
6. Being HIV negative
7. Without any cardiovascular disease
8. Being active in sex work (for the Female commercial sex worker group)

Exclusion criteria:

1. Age less than 18 years or more than 50 years old
2. Pregnancy (if a women becomes pregnant during the 10 weeks of the project she will be excluded)
3. Breast feeding
4. Pregnant in the last 12 months
5. Being positive for Sexual transmissible disease or bacterial vaginosis at week 0
6. Menopausal
7. No longer involve in sex work (for the female sex worker group)
8. Having a chronic disease
9. Taking any of the medication listed in annex 1 for health conditions
10. Being allergic to acetylsalicylic acid, other medication for pain or fever, tartrazine dye or chloroquine, hydroxuchloroquine, primaquine or any other medication
11. Having heartburn, stomach pain, stomach ulcer, anemia, hemophilia, kidney or liver disease, psoriasis, porphyria or other blood disease, G-6-PD deficiency, dermatitis (skin inflammation), alcoholism
12. Having experienced previous vision changes while taking chloroquine, hydroxychloroquine (Aralen) or primaquine.
13. Having a history of a diagnosed cardiovascular event, heart failure, peripheral arterial disease, angina, stoke, transient ischemic attack
14. Having a current or recurrent condition with a high risk of major bleeding
15. Having anemia
16. Current participation in a clinical trial

    -

    -

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 91 (Actual)
Dates: Start 2014-04; Primary Completion 2015-12 (Actual); Study Completion 2018-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith R. Fowke, PhD, Principal Investigator — University of Manitoba
Locations (1):
- Kenyan Aids Control Project/University of Nairobi, Nairobi, Kenya

REFERENCES:
- [Derived] Lajoie J, Kowatsch MM, Mwangi LW, Boily-Larouche G, Oyugi J, Chen Y, Kimani M, Ho EA, Kimani J, Fowke KR. Low-Dose Acetylsalicylic Acid Reduces T Cell Immune Activation: Potential Implications for HIV Prevention. Front Immunol. 2021 Nov 18;12:778455. doi: 10.3389/fimmu.2021.778455. eCollection 2021. PMID 34868050
- [Derived] Lajoie J, Mwangi L, Fowke KR. Preventing HIV infection without targeting the virus: how reducing HIV target cells at the genital tract is a new approach to HIV prevention. AIDS Res Ther. 2017 Sep 12;14(1):46. doi: 10.1186/s12981-017-0166-7. PMID 28893304

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Acetylsalicylic Acid (ASA) | Hydroxychloroquine (HCQ)
Started | 43 | 48
Completed | 37 | 39
Not Completed | 6 | 9
Not completed — Lost to Follow-up | 5 | 7
Not completed — Became STIs Positive | 1 | 2

BASELINE CHARACTERISTICS:
Population: study population was women from the general population in general good health and HIV negative
Groups:
- Total: Total of all reporting groups
Arm/Group | Acetylsalicylic Acid (ASA) | Hydroxychloroquine (HCQ) | Total
Number analyzed (Participants) | 43 | 48 | 91
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 43 | 48 | 91
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 48 | 91
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Kenya | 43 | 48 | 91
T cell immune activation [Mean (Standard Deviation); unit: percentage of cells] | 30.82 (20.08) | 30.49 (14.34) | 30.64 (15.06)

OUTCOME MEASURES:

1. Primary Outcome: Changes in Systemic Immune Activation From Baseline Observed by the CD69 Expression on CD4 T Cells
Description: We will analyse reduce of immune activation by measuring change in T cell activation (CD69) between baseline and every month during drug administration phase (8 weeks).
Time Frame: Baseline and 8 weeks
Population: general population
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Acetylsalicylic Acid (ASA) | Hydroxychloroquine (HCQ)
Number analyzed (Participants) | 43 | 48
percentage of cells
  Average of CD4+CD69+ at baseline | 4.04 (3.83) | 5.55 (5.09)
  Average of CD4+CD69+ T cells cells after treatment | 4.9 (4.4) | 4.99 (3.56)

2. Secondary Outcome: Change in Number of CCR5+CD4+ T Cell Population at the Female Genital Tract.
Description: We will measure changes in the number of CD4+T cells expressing CCR5 at the female genital tract before and at the end of the study.
Time Frame: baseline and 8 weeks
Measure: Median (Standard Deviation); unit: percentage of cells
Arm/Group | Acetylsalicylic Acid (ASA) | Hydroxychloroquine (HCQ)
Number analyzed (Participants) | 43 | 48
percentage of cells | 17.60 (11.27) | 22.10 (14.93)

ADVERSE EVENTS:
Arm/Group | Acetylsalicylic Acid (ASA) | Hydroxychloroquine (HCQ)
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/48
Other Adverse Events (participants affected / at risk) | 0/43 | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No